CLINICAL TRIAL: NCT00443248
Title: A 2-Way Repeatability Study To Investigate Vaginal Blood Flow Before, During And After Visual Sexual Stimulation In Pre- And Post-Menopausal Women With And Without Female Sexual Arousal Disorder, Using The Heat Wash-Out Technique.
Brief Title: Vaginal Heat Wash-out (HWO) in 4 Groups of Women (Pre- and Postmenopausal With and Without Female Sexual Arousal Disorder (FSAD)).
Acronym: FSAD HWO VBF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A9001302
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Sexual Dysfunction, Physiological
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaginal Heat Wash-Out Device (Experimental)
  Interventions: Device: Vaginal Heat Wash-Out Device

INTERVENTIONS:
Device: Vaginal Heat Wash-Out Device — No drug administered. Device tested twice with each subject.

SUMMARY:
The Pfizer developed Heat Wash-Out (HWO) system is a software controlled electromechanical system designed to measure vaginal wall blood flow. A small vaginal probe is attached to a control unit. Output data are collected on a PC. By measuring the clearance of heat from the heated probe, a direct measure of absolute blood flow can be obtained. The study will assess the technique's ability to differentiate between pre- and post-menopausal women; with and without Female Sexual Arousal Disorder (FSAD).

DETAILED DESCRIPTION:
Medical Device Development

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women aged 18-40 (with and without FSAD) or
* Post-menopausal women aged 50-65 (with and without FSAD.
* FSAD must have been present for at least 6 months.

Exclusion Criteria:

* Pregnant or lactating women (pre-menopausal population)
* Systemic Hormone Replacement Therapy (HRT) or Selective Estrogen Receptor Modulator (SERM) (postmenopausal population)
* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic disease or other major psychological or sexual disorder.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To assess the safety and toleration of the heat washout device. | 2 weeks
To investigate differences in vaginal blood flow following visual sexual stimulation in pre-menopausal women with and without FSAD. | 2 weeks

SECONDARY OUTCOMES:
To investigate changes in subjective acute sexual arousal following visual sexual stimulation in women with and without FSAD. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Australia (2):
  - Pfizer Investigational Site, Dulwich, South Australia
  - Pfizer Investigational Site, Nedlands, Western Australia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001302